CLINICAL TRIAL: NCT06451861
Title: Randomized Study of ABC-14 Regimen ( AZA, Venetoclax and Chidamide) Compared With "3+7" Standard Induction Therapy or AB-14 (Venetoclax Combined With Azacitidine) for Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Randomized Study of ABC-14 Regimen Compared With "3+7" Standard Induction Therapy or AB-14 for ND AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABC-14_101
Record Dates: First submitted 2024-02-05; First posted 2024-06-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: ABC-14 regimen; "3+7" regimen; AB-14 regimen
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; venetoclax; Azacitidine; Anthracyclines; Anthraquinones; Idarubicin; Daunorubicin; Mitoxantrone; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABC-14 regimen (Experimental): AZA,Venetoclax,Chidamide
  Interventions: Drug: Chidamide; Drug: Venetoclax; Drug: azacitidine
- 3+7 chemotherapy regimen (Active Comparator): Daunorubicin/idarubicin/mitoxantrone and cytarabine
  Interventions: Drug: Anthracyclines or anthraquinones; Drug: cytarabine
- AB-14 regimen (Active Comparator): AZA,Venetoclax
  Interventions: Drug: Venetoclax; Drug: azacitidine

INTERVENTIONS:
Drug: Chidamide — Induction Therapy
  Arms: ABC-14 regimen
Drug: Venetoclax — Induction Therapy
  Arms: AB-14 regimen; ABC-14 regimen
Drug: azacitidine — Induction Therapy
  Arms: AB-14 regimen; ABC-14 regimen
Drug: Anthracyclines or anthraquinones — Induction Therapy
  Other Names: idarubicin; daunorubicin; mitoxantrone
  Arms: 3+7 chemotherapy regimen
Drug: cytarabine — Induction Therapy
  Arms: 3+7 chemotherapy regimen

SUMMARY:
To compare the efficacy and safty of ABC-14 regimen with the traditional "3+7" regimen or AB-14 regimen in the treatment of newly diagnosed acute myeloid leukaemia

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a clonal malignant blood disease with genetic heterogeneity and originated from hematopoietic stem progenitor cells.In the past 50 years, the "3+7" induction regimen represented by cytotoxic drugs (including anthracyclines/anthraquinones combined with cytarabine) has remained the standard induction regimen for newly diagnosed AML patients with intensive chemotherapy. In AML patients <60 years old, the "3+7" regimen induces a complete response rate of 60% to 80%, but the treatment-related mortality is as high as 13%, and more than half of the patients face the threat of relapse, and the 5-year overall survival rate is about 35% to 40%.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with AML (the diagnostic criteria refer to WHO2022 standard, non-APL), and have not received systemic anti-leukemia therapy (except hydroxyurea, low-dose cytarabine and other tumor reduction pretreatments);
2. Age ≥18 years old;
3. ECOG≤4;
4. The fertile woman agrees to use effective contraception during the treatment period and up to 3 months after the end of the treatment; Sign the informed consent form.

Exclusion Criteria:

1. Known history of allergy to the investigational drug;
2. Resistance to azacytidine, azacitidine, Venetoclax;
3. Inability to take oral medication;
4. Combined with uncontrolled active infections (including bacterial, fungal or viral infections);
5. Combined with uncontrolled major organ dysfunction: cardiac insufficiency, decompensated liver insufficiency, moderate/severe renal insufficiency, etc.;
6. Participating in other clinical studies that affect the main purpose of this study; Patients deemed unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission (CRc) | 2 months
  composite complete remission，CRc: CR + CRi + MLFS

SECONDARY OUTCOMES:
the rate of MRD turn negative | 6 months
  minimal residual disease turn negative
DoR | 2 year
  Duration of remission
RFS | 1 year
  Relapsed-free survival
OS | 1 year
  Overall survival
AE | Throughout the study until the end, up to 2 years
  Incidence of of grade 3-4 adverse events/Duration of severe myelosuppression/ Incidence of severe infection/Treatment-related mortality, according to Common Terminology Criteria for Adverse Events, versions 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jianyu Weng, Principal Investigator — Guangdong Provincial People Hosptial
Locations (13):
- China (13):
  - Dongguan General Hosptial, Dongguan, Guangdong
  - Foshan First People's Hospital, Foshan, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen second people's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Zhuhai General Hosptial, Zhuhai, Guangdong
  - Hainan General Hosptial, Haikou, Hainan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan H, Huang X, Wu P, Deng C, Li M, Lai P, Du X, Weng J. Comparing the efficacy and safety of the ABC-14 regimen (azacitidine, venetoclax, and chidamide) with traditional "3 + 7" intensive induction regimen or AB-14 regimen (venetoclax combined with azacitidine) in newly diagnosed AML: study protocol for a prospective, multicenter, randomized, open-label clinical trial. Trials. 2025 Dec 10;27(1):38. doi: 10.1186/s13063-025-09339-y. PMID 41366419